CLINICAL TRIAL: NCT04638023
Title: Arabin Pessary Use in Women at High Risk for Preterm Birth: 7 Years' Experience in a Single Tertiary Centre
Brief Title: Arabin Pessary in Singleton Pregnancy
Status: Completed | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Assoc. Prof., National University of Malaysia
Other Study IDs: FF-2017-372
Record Dates: First submitted 2020-11-15; First posted 2020-11-20 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Previous Mid Trimester Miscarriage; Previous Preterm Birth; Previous Cervical Surgery; Short Cervix on Ultrasound
Keywords: Arabin pessary, spontaneous preterm birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Arabin pessary — Arabin pessary was inserted intravaginally electively in women with cervical insufficiency (history based) or as emergency in those with short cervix on ultrasound.

SUMMARY:
This was a retrospective study sharing the experience of women high risk for spontaneous preterm birth managed by Arabin pessary.

DETAILED DESCRIPTION:
The study recruitment was from 1st January 2013 until 31st December 2019. Inclusion criteria were previous mid-trimester miscarriage and/or preterm birth, previous cervical surgery or short cervical length on routine ultrasound. The primary outcome measure was birth before 34 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* all women high risk for spontaneous preterm birth

Exclusion Criteria:

* had Arabin insertion elsewhere
* delivered elsewhere
* incomplete record

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Study Population: All women high risk for spontaneous preterm birth who were managed with Arabin pessary were included.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Birth at or more than 34 weeks | From insertion of the Arabin pessary until birth of the foetus
  Gestation of birth in percentage that occurred at or more than 34 weeks gestation

SECONDARY OUTCOMES:
Type of labour | From insertion of the Arabin pessary until birth of the foetus
  Type of labour whether spontaneous or induced
Mode of delivery | From onset of labour until birth of the foetus
  Mode of delivery whether vaginal or caesarean section
Median birth weight | At birth
  Median neonatal birth weight in gram
Admission into neonatal intensive care unit | At birth until discharged from the hospital
  The need to admit the neonate to neonatal care intensive care unit at birth
Mean cervical length | At insertion of the Arabin pessary
  The mean cervical length at insertion of the Arabin pessary
Subsequent management | From insertion of Arabin pessary until birth of the foetus
  The management of the patients after insertion of the Arabin pessary
Combination with progestogen therapy | from insertion of Arabin pessary until birth of the foetus
  Addition of progestogen therapy either vaginally or parenterally
Complications | From insertion of Arabin pessary until birth of the foetus
  Antenatal complications such as diabetes, hypertension and rupture of membranes

CONTACTS AND LOCATIONS:
Overall Officials: Rahana Abd Rahman, Principal Investigator — UKM
Locations (1):
- National University of Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Methodology

REFERENCES:
- [Derived] Rahman RA, Atan IK, Ali A, Kalok AM, Ismail NAM, Mahdy ZA, Ahmad S. Use of the Arabin pessary in women at high risk for preterm birth: long-term experience at a single tertiary center in Malaysia. BMC Pregnancy Childbirth. 2021 May 10;21(1):368. doi: 10.1186/s12884-021-03838-x. PMID 33971828